CLINICAL TRIAL: NCT06922760
Title: Utilizing CT Based Imaging Parameters of Body Composition to Understand Heterogeneity of Response to Biologic Therapies in Severe Asthma Cohorts
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Njira Lugogo, Associate Professor of Internal Medicine, University of Michigan
Other Study IDs: HUM00140217
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- University of Michigan, Ann Arbor, MI: Severe asthma patients treated at Michigan Medicine who are on biologic therapies for asthma and who have CT imaging and known outcomes on therapy.
  No interventions were included in this retrospective study.
- National Jewish Health, Denver, CO: Severe asthma patients treated at National Jewish Health who are on biologic therapies for asthma and who have CT imaging and known outcomes on therapy.
  No interventions were included in this retrospective study.

SUMMARY:
This study will utilize University of Michigan EMR data to form a retrospective cohort of severe asthma patients on biologic therapies for asthma with computed tomography (CT) imaging and known outcomes on therapy. These images will then be analyzed using morphomics, a combination of high-throughput image analysis and deep learning techniques, to derive imaging biomarkers that will be able to predict therapeutic response to biologics. These biomarkers will then be tested in a second cohort from the National Jewish Health to assess for validity.

DETAILED DESCRIPTION:
The two arms for this study represent the two cohorts: the University of Michigan cohort, and the National Jewish Health cohort. The cohorts were split into arms, as the National Jewish Health cohort was intended to act as a validator group for results derived from participants in the University of Michigan cohort.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosis defined as a positive methacholine test, supportive PFTs, or clinician diagnosis with appropriate supporting clinical context
* Prescribed and taking an FDA-approved biologic medication for severe asthma (mepolizumab, benralizumab, reslizumab, omalizumab, or dupilumab)
* Chest computerized tomography (CT) images taken for any clinical purpose

Exclusion Criteria:

* 10-year history of smoking
* Evidence of emphysema on CT imaging
* Severe bronchiectasis secondary to other causes (subjects with scattered bronchiectasis secondary to severe asthma will not excluded)
* Lack of accessible adequate follow-up information (4 or more months from drug initiation with clear documentation of response) will be excluded from final analysis due to inability to assess response but will be included in the initial cluster identification

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 500 male or female subjects ages 18-85 with a diagnosis of asthma, on biologic therapy , and with a pre-biologic CT scan for any clinical purpose drawn from Michigan Medicine EHR (University of Michigan in Ann Arbor, MI, USA) and National Jewish Health (Denver, Colorado, USA).
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Njira Lugogo, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - National Jewish Health, Denver, Colorado
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | University of Michigan, Ann Arbor, MI | National Jewish Health, Denver, CO
Started | 152 | 81
Completed | 152 | 81
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | University of Michigan, Ann Arbor, MI | National Jewish Health, Denver, CO | Total
Number analyzed (Participants) | 152 | 81 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.39 (14.31) | 51.75 (15.58) | 52.17 (14.73)
Age, Customized [Mean (Standard Deviation); unit: years] — Population: Data is the specific breakdown of mean participant age by gender.
  years
    Female: number analyzed (Participants) | 105 | 40 | 145
    Female | 51.42 (13.21) | 48.08 (17.86) | 50.50 (14.65)
    Male: number analyzed (Participants) | 47 | 41 | 88
    Male | 54.55 (16.46) | 55.34 (12.15) | 54.92 (14.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 40 | 145
  Male | 47 | 41 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 12 | 15
  Not Hispanic or Latino | 144 | 68 | 212
  Unknown or Not Reported | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 2 | 23
  White | 125 | 69 | 194
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 10 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 152 | 81 | 233
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Data is the specific breakdown of mean participant BMI by gender.
  kg/m^2
    Female: number analyzed (Participants) | 105 | 40 | 145
    Female | 32.46 (9.27) | 31.70 (9.21) | 32.25 (9.23)
    Male: number analyzed (Participants) | 47 | 41 | 88
    Male | 29.97 (4.92) | 30.62 (5.61) | 30.27 (5.23)
Height [Mean (Standard Deviation); unit: centimeters] — Population: Data is the specific breakdown of mean participant height by gender.
  centimeters
    Female: number analyzed (Participants) | 105 | 40 | 145
    Female | 162.31 (6.78) | 162.84 (6.05) | 162.45 (6.57)
    Male: number analyzed (Participants) | 47 | 41 | 88
    Male | 176.95 (6.56) | 176.59 (7.78) | 176.78 (7.12)
Weight [Mean (Standard Deviation); unit: kilograms] — Population: Data is the specific breakdown of mean participant weight by gender.
  kilograms
    Female: number analyzed (Participants) | 105 | 40 | 145
    Female | 85.31 (23.83) | 83.85 (23.89) | 84.91 (23.77)
    Male: number analyzed (Participants) | 47 | 41 | 88
    Male | 93.99 (16.88) | 95.43 (18.33) | 94.66 (17.48)

OUTCOME MEASURES:

1. Primary Outcome: Chest Wall Muscle Size
Description: Muscle size was measured as the skeletal muscle cross-sectional area in centimeters squared (cm2) measured at the level of the T10 vertebra to determine the cutoff value in chest wall muscle size that optimally classified patients that had and did not have any reduction in pre-treatment baseline exacerbation frequency (binary).
Time Frame: 28 months
Population: 8 participants in the University of Michigan arm and 1 participant in the National Jewish Health arm did not have either a baseline or post-treatment count of exacerbations so the outcome could not be computed for them. In addition, 20 participants in the National Jewish Health arm (including the 1 without complete outcome data) did not have complete skeletal muscle visible within the scan field, so muscle size and quality could not be adequately assessed.
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | University of Michigan, Ann Arbor, MI | National Jewish Health, Denver, CO
Number analyzed (Participants) | 144 | 61
cm2
  Had reduction in exacerbations: number analyzed (Participants) | 122 | 43
  Had reduction in exacerbations | 95.49 (25.63) | 97.82 (29.04)
  Did not have reduction in exacerbations: number analyzed (Participants) | 22 | 18
  Did not have reduction in exacerbations | 87.98 (23.65) | 102.86 (28.77)

2. Primary Outcome: Chest Wall Muscle Quality
Description: Muscle quality was measured as the skeletal muscle density in Hounsfield Units (HU) to determine the cutoff value in chest wall muscle quality that optimally classified patients that had and did not have any reduction in pre-treatment baseline exacerbation frequency (binary).
Time Frame: 28 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: HU
Arm/Group | University of Michigan, Ann Arbor, MI | National Jewish Health, Denver, CO
Number analyzed (Participants) | 144 | 61
HU
  Had a reduction in exacerbations: number analyzed (Participants) | 122 | 43
  Had a reduction in exacerbations | 36.57 (7.94) | 30.27 (7.28)
  Did not have reduction in exacerbations: number analyzed (Participants) | 22 | 18
  Did not have reduction in exacerbations | 39.18 (6.96) | 28.60 (6.43)

3. Primary Outcome: Exacerbation Reduction - Muscle Size
Description: Muscle size was measured as the skeletal muscle cross-sectional area in centimeters squared (cm2) measured at the level of the T10 vertebra to assess whether skeletal muscle size area could be used to predict exacerbation frequency. Results reflect the average muscle sizes when frequency could be predicted.
Time Frame: 28 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | University of Michigan, Ann Arbor, MI | National Jewish Health, Denver, CO
Number analyzed (Participants) | 144 | 61
cm2 | 94.3 (25.4) | 99.3 (28.8)
Statistical Analysis 1: Comparison: University of Michigan, Ann Arbor, MI; Test type: Other — Statistical Test of Hypothesis; p = 0.411, Regression, Linear
Statistical Analysis 2: Comparison: National Jewish Health, Denver, CO; Test type: Other — Statistical Test of Hypothesis; p = 0.161, Regression, Linear

4. Primary Outcome: Exacerbation Reduction - Muscle Quality
Description: Muscle quality was measured as the skeletal muscle density in Hounsfield Units (HU) to determine the cutoff value in chest wall muscle quality to assess whether skeletal muscle quality could be used to predict exacerbation frequency. Results reflect the average muscle sizes when frequency could be predicted.
Time Frame: 28 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: HU
Arm/Group | University of Michigan, Ann Arbor, MI | National Jewish Health, Denver, CO
Number analyzed (Participants) | 144 | 61
HU | 37 (7.8) | 29.8 (7)
Statistical Analysis 1: Comparison: University of Michigan, Ann Arbor, MI; Test type: Other — Statistical Test of Hypothesis; p = 0.007, Regression, Linear
Statistical Analysis 2: Comparison: National Jewish Health, Denver, CO; Test type: Other — Statistical Test of Hypothesis; p = 0.5, Regression, Linear

5. Primary Outcome: Exacerbations
Description: The number of exacerbations post-biologic were compared to the the number of baseline exacerbations. Baseline measurements were counted in the year prior to biologic initiation. Any exacerbation recorded between 4 to 28 months after biologic initiation was recorded as a post-biologic exacerbation. Any reduction in between the pre- and post-biologic was counted as an exacerbation reduction. Results reflect the number of participants who experienced (True) or did not experience (False) a reduction in exacerbations.
Time Frame: pre-biologic at baseline (looking back 1 year), post-biologic (4-18 months after biologic)
Population: 8 participants in the University of Michigan arm and 1 participant in the National Jewish Health arm did not have either a baseline or post-treatment count of exacerbations so the outcome could not be computed for them.
Measure: Count of Participants; unit: Participants
Arm/Group | University of Michigan, Ann Arbor, MI | National Jewish Health, Denver, CO
Number analyzed (Participants) | 144 | 80
Participants
  True | 122 | 61
  False | 22 | 19

6. Secondary Outcome: FEV1 Improvement
Description: Muscle size was used to investigate body composition measures associated with a 5% or greater improvement in forced expiratory volume in one second (FEV1). Muscle size was measured as the skeletal muscle cross-sectional area in centimeters squared (cm2) measured at the level of the T10 vertebra to determine the cutoff value in chest wall muscle size that optimally classified participants who had and did not have improvement in FEV1. Participants with ≥5% improvement in FEV1 during the 4 to 18-month period following initiation of biologics were classified as responders. Any participant who did not achieve a ≥5% improvement from baseline in that timeframe was classified as a non-responder.
Time Frame: pre-biologic at baseline (looking back 1 year), post-biologic (4-18 months after biologic)
Population: 48 UM patients and 31 NJ patients that lacked a suitable CT and pre- and post-biologic FEV1 measure were not included in this analysis
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | University of Michigan, Ann Arbor, MI | National Jewish Health, Denver, CO
Number analyzed (Participants) | 104 | 50
cm2
  Responders: number analyzed (Participants) | 46 | 25
  Responders | 94.59 (25.06) | 96.93 (32.43)
  Non-Responders: number analyzed (Participants) | 58 | 25
  Non-Responders | 88.31 (23.85) | 102.81 (25.26)

7. Secondary Outcome: Reduction in Oral Corticosteroid (OCS)
Description: Muscle size was used to investigate body composition measures associated with any reduction in maintenance OCS use when compared to baseline OCS use. Subjects with any OCS reduction in use during the 4- to 18-month period following initiation of biologics were classified as responders.
Time Frame: pre-biologic at baseline (looking back 1 year), post-biologic (4-18 months after biologic)
Population: 25 UM patients and 20 NJ patients that lacked a suitable CT and pre- and post-biologic OCS maintenance use were not included in this analysis
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | University of Michigan, Ann Arbor, MI | National Jewish Health, Denver, CO
Number analyzed (Participants) | 127 | 61
cm2
  Responders: number analyzed (Participants) | 33 | 14
  Responders | 91.17 (23.84) | 103.94 (32.96)
  Non-Responders: number analyzed (Participants) | 94 | 47
  Non-Responders | 96.09 (26.17) | 97.92 (27.71)

ADVERSE EVENTS:
Description: Adverse event data was not collected, as this was a retrospective observational study.
Arm/Group | University of Michigan, Ann Arbor, MI | National Jewish Health, Denver, CO
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT06922760/Prot_SAP_000.pdf